CLINICAL TRIAL: NCT05349175
Title: Augmented Infant Resuscitator (AIR): Transitioning a Novel Behavior Change Innovation to Drive Newborn Ventilation Skills Enhancement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Grand Challenges Canada (Other)
Responsible Party: Principal Investigator, Brett D. Nelson, MD, MPH, DTM&H, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2013P002204b
Record Dates: First submitted 2022-04-15; First posted 2022-04-27 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Asphyxia Neonatorum; Birth Asphyxia; Perinatal Asphyxia
MeSH Terms: conditions — Asphyxia Neonatorum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): Receives AIR device feedback beginning immediately after training
  Interventions: Device: Augmented Infant Resuscitator (AIR)
- Cohort B (Experimental): Receives AIR device feedback beginning 2 months after training
  Interventions: Device: Augmented Infant Resuscitator (AIR)
- Cohort C (Experimental): Receives AIR device feedback beginning 4 months after training
  Interventions: Device: Augmented Infant Resuscitator (AIR)

INTERVENTIONS:
Device: Augmented Infant Resuscitator (AIR) — Real-time visual feedback from the AIR device regarding quality of bag-mask ventilation

SUMMARY:
Augmented Infant Resuscitator (AIR) is an inexpensive add-on, compatible with nearly every existing bag-valve mask and many types of ventilation equipment. AIR monitors ventilation quality and provides real-time objective feedback and actionable cues to clinicians to both shorten training times and improve resuscitation quality, adoption, retention, and confidence.

DETAILED DESCRIPTION:
The investigators propose a randomized controlled trial to asses the impact, feasibility, and acceptability of real-time visual feedback from the AIR device. The study will begin by training and equipping all available skilled birth attendants (SBAs) at the participating facilities in the Helping Babies Breathe (HBB) training curriculum. SBAs will also receive HBB Provider Guides and wall-mountable HBB action plans. Immediately before and after training, the study teams will use the traditional HBB assessment tools to evaluate SBAs' HBB knowledge and skills.

Facilities will then be randomized, by cluster, to either receive AIR feedback at the start of the trial (Cohort A) or beginning at 2 (Cohort B) or 4 months post-training (Cohort C). Both intervention and control cohorts will be encouraged to start regular "low-dose, high-frequency" (LDHF) practice with the AIR devices. LDHF involves frequent "doses" of shorter, often skills- or competency-based, individual- or pair-learning practice sessions. Study teams will establish HBB practice corners in each health facility, consisting of HBB equipment, NeoNatalie, AIR device, HBB Action Plan, and a log book.

Participants in Cohort A will practice with AIR devices providing visual feedback immediately post-training, while Cohorts B and C will start with AIR devices without visual feedback. Disabling feedback from the device does not compromise its recording function that collects time-stamped data on ventilation quality. Cohort B will switch to AIR device feedback at 2 months, and Cohort C will switch to AIR device feedback at 4 months. All cohorts will continue LDHF practice with AIR device feedback through up to 6 months after initial HBB training.

During the study, the study teams will conduct facility-based bag-mask ventilation (BMV) assessments at 2, 4, and 6 months. The primary outcome for this measurement will be duration of effective ventilation in a two-minute window after initiation of ventilation, as part of the HBB program's existing BMV skills check and OSCE B. "Effective ventilation" is defined as ventilating in the correct rate range without airway blockages, significant leaks, and harsh breaths and will be determined by the AIR device. Note, during these skills assessments, study participants will be evaluated with feedback turned off during the two-minute breathing epoch.

After AIR feedback is turned on at a facility, de-identified device-recorded data on provider-level frequency and quality of practice will be aggregated, shared, and discussed with each health center every 2 months to support and harmonize with their existing facility-led quality improvement efforts.

ELIGIBILITY:
Inclusion Criteria:

* Skilled birth attendants (SBAs) working clinically at the selected facilities (i.e., in-service providers)
* SBAs who participate in the HBB training offered by our group at the beginning of the study
* SBAs who demonstrate competence, after initial training, in key neonatal resuscitation skills and competencies (i.e., pass the BMV skills check and OSCE B)
* SBAs able to adequately understand the language in which the HBB training is offered (e.g., the investigators anticipate the trainings will be offered in English)
* SBAs over 18 years of age
* SBAs who provide written informed consent for participation in the study

Exclusion Criteria:

* Students or clinicians still in training (i.e., pre-service providers)
* SBAs and other health workers who do not participate in initial HBB training
* SBAs that are unable to adequately understand the language in which the HBB training is offered
* SBAs under 18 years of age
* SBAs who do not provide written informed consent for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Effective bag-mask ventilation | 2 minutes
  Duration of effective bag-mask ventilation by clinician during a 2-minute trial. This is measured internally from the AIR device. "Effective ventilation" is defined as having all three of the following conditions simultaneously: (1) Correct rate (30-60 breaths per minute); (2) Absence of significant leak (compliance >4.0mL/cm H2O); and (3) Absence of a significant airway blockage (defined as compliance <0.10 mL/cm H2O or resistance >90 cmH2O/L/s). These measurements are determined by sensors in the AIR device for all arms of the study. Their accuracy for manikin use was determined to be 100% in the following trial: Bennett el al. Anesth Analgesia. 2018 Mar;126(3):947-955. doi: 10.1213/ANE.0000000000002432.
Time to effective bag-mask ventilation | 2 minutes
  How long it takes for clinician to achieve effective ventilation during 2-minute trial -- timed from when the mask first touches the face of the manikin until all three icons are green. This is measured by an observer using a stop-watch. Again, "effective ventilation" is defined as having all three of the following conditions simultaneously and is indicated to the RA by all three icons on the AIR device turning green: (1) Correct rate (30-60 breaths per minute); (2) Absence of significant leak (compliance >4.0mL/cm H2O); and (3) Absence of a significant airway blockage (defined as compliance <0.10 mL/cm H2O or resistance >90 cmH2O/L/s).
Bag-mask ventilation skills immediately after training | Immediately after training
  Clinicians' bag-mask ventilation skills will be assessed immediately after training. Assessment of these skills will be done using current standards, namely the HBB program's 'Bag-mask ventilation skills test' and 'OSCE B.'
Bag-mask ventilation skills 2 months post-training | 2 months after training
  Clinicians' bag-mask ventilation skills will be assessed 2 months after training. Assessment of these skills will be done using current standards, namely the HBB program's 'Bag-mask ventilation skills test' and 'OSCE B.'
Bag-mask ventilation skills 4 months post-training | 4 months after training
  Clinicians' bag-mask ventilation skills will be assessed 4 months after training. Assessment of these skills will be done using current standards, namely the HBB program's 'Bag-mask ventilation skills test' and 'OSCE B.'
Bag-mask ventilation skills 6 months post-training | 6 months after training
  Clinicians' bag-mask ventilation skills will be assessed 6 months after training. Assessment of these skills will be done using current standards, namely the HBB program's 'Bag-mask ventilation skills test' and 'OSCE B.'

SECONDARY OUTCOMES:
Provider-level perceptions - focus groups | 6 months
  Provider perceptions of the AIR device, using focus group discussions.
Provider-level perceptions - interviews | 6 months
  Provider perceptions of the AIR device, using semi-structured interviews.
Cost analysis | 6 months
  Cost analysis for implementation and evaluation of the AIR device

CONTACTS AND LOCATIONS:
Overall Officials: Brett D. Nelson, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bennett DJ, Itagaki T, Chenelle CT, Bittner EA, Kacmarek RM. Evaluation of the Augmented Infant Resuscitator: A Monitoring Device for Neonatal Bag-Valve-Mask Resuscitation. Anesth Analg. 2018 Mar;126(3):947-955. doi: 10.1213/ANE.0000000000002432. PMID 28863023
- [Result] Ali A, Nudel J, Heberle CR, Santorino D, Olson KR, Hur C. Cost effectiveness of a novel device for improving resuscitation of apneic newborns. BMC Pediatr. 2020 Jan 30;20(1):46. doi: 10.1186/s12887-020-1925-5. PMID 32000740